CLINICAL TRIAL: NCT01347099
Title: Internet-based Cognitive Behavior Therapy for Obsessive Compulsive Disorder: A Randomized Controlled Trial
Brief Title: Internet-based Cognitive Behavior Therapy (CBT) for Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Nils Lindefors, Psykiatri Sydväst
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCD-S
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2011-05

CONDITIONS: Obsessive Compulsive Disorder
Keywords: CBT; OCD; Internet; Reduce symptom burden
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet CBT (Experimental): Internet-delivered CBT. Contact with therapist thru an e-mail system. 10 weeks.
  Interventions: Behavioral: Internet-based cognitive behavior therapy
- Support therapy (Placebo Comparator): 10 weeks. Therapist support contact through e-mail.
  Interventions: Behavioral: Support therapy on Internet

INTERVENTIONS:
Behavioral: Internet-based cognitive behavior therapy — Internet-delivered CBT. Contact with therapist thru an e-mail system. 10 weeks
  Arms: Internet CBT
Behavioral: Support therapy on Internet — Internet-delivered support therapy. Contact with therapist thru an e-mail system. 10 weeks
  Arms: Support therapy

SUMMARY:
Cognitive behavior therapy (CBT) is an effective treatment for obsessive compulsive disorder (OCD) but there is a lack of properly trained CBT therapists. One possible treatment alternative is Internet-based CBT (ICBT) with minimal therapist input. The aim of this study was therefore to evaluate ICBT for OCD.

DETAILED DESCRIPTION:
This is a randomized controlled trial with 101 participants. The control group receives support therapy on demand on the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of obsessive compulsive disorder (OCD)
* At least 18 years old
* Able to read and write in swedish
* Computer access

Exclusion Criteria:

* other primary diagnosis
* substance abuse,
* psychosis,
* bipolar disorder,
* suicidal ideation,
* adjusted pharmacological treatment the last two months
* current psychological treatment for OCD,
* been treated with CBT the last two years,
* serious somatic disease,
* Y---BOCS>31
* hoarding as primary OCD subtype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06

PRIMARY OUTCOMES:
Change from Baseline of obsessions and compulsions after 10 weeks and at 3- and 12 months after treatment. | Two weeks before treatment, 10 weeks after treatment starts, 3 and 12 months after treatment has ended
  Yale Brown Obsessive Compulsive Scale (Y-BOCS)

SECONDARY OUTCOMES:
Change from Baseline of obsessions and compulsions after 10 weeks and at 3- and 12 months after treatment. | Two days before treatment, once per week for 10 weeks after treatment starts, 3 and 12 months after treatment has ended
  Obsessive Compulsive Scale - Revised (OCI-R)
Change from Baseline of obsessions and compulsions after 10 weeks and at 3- and 12 months after treatment. | Two weeks before treatment, 10 weeks after treatment starts, 3 and 12 months after the treatment has ended
  Dimensional Obsessive Compulsive Scale (DOCS)
Change from Baseline of depressive symptoms after 10 weeks and at 3- and 12 months after treatment. | Two weeks before treatment, 10 weeks after treatment starts, 3 and 12 months after treatment has ended
  Montgomery Asberg Depression Rating Scale
Change from Baseline of meta cognitions after 10 weeks and at 3- and 12 months after treatment. | Two weeks before treatment, 10 weeks after treatment starts, 3 and 12 months after treatment has ended
  Obsessive Beliefs Scale
Change from Baseline of quality of life after 10 weeks and at 3- and 12 months after treatment. | Two weeks before treatment, 10 weeks after treatment starts, 3 and 12 months after treatment has ended
  Euroqol

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, MD, PhD, Principal Investigator — Department of Clinical Neuroscience, KI
Locations (1):
- Psykiatri Sydväst, Stockholm, Sweden

REFERENCES:
- [Result] Andersson E, Enander J, Andren P, Hedman E, Ljotsson B, Hursti T, Bergstrom J, Kaldo V, Lindefors N, Andersson G, Ruck C. Internet-based cognitive behaviour therapy for obsessive-compulsive disorder: a randomized controlled trial. Psychol Med. 2012 Oct;42(10):2193-203. doi: 10.1017/S0033291712000244. Epub 2012 Feb 21. PMID 22348650